CLINICAL TRIAL: NCT05121220
Title: Efficacy and Cost-effectiveness of Orthodontic Retention Protocols
Acronym: orthoretenti
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poliklinika Orthonova (Other)
Collaborators: University of Zagreb School of Dental Medicine, Zagreb, Croatia (Unknown); University of Rijeka Faculty of Dental Medicine, Rijeka, Croatia (Unknown)
Responsible Party: Principal Investigator, silvija kanižaj ugrin, Dentist, Orthodontic specialist, Poliklinika Orthonova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 66771011
Record Dates: First submitted 2021-10-02; First posted 2021-11-16 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Orthodontic Relapse
Keywords: retention wire; fixed retainer; orthodontic therapy
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fixed mandibular lingual rectangular retainer 0.673 x 0.268 mm (Experimental): 0.673 x 0.268 mm 8-stranded wire Bond A Braid (Reliance Orthodontic Products, USA) will be bonded in mandible canine to canine on each tooth using Filtek flowable composite (Ivoclar Vivadent, Lichtenstein) and Multilink adhesive (3M, USA).
  Interventions: Device: fixed retainer
- fixed mandibular lingual round retainer 0.40 mm (Experimental): 0.40 mm round 6-stranded wire (Forestadent, Germany) will be bonded on 6 mandibular frontal teeth, canine to canine on each tooth using Filtek flowable composite (Ivoclar Vivadent, Lichtenstein) and Multilink adhesive (3M, USA).
  Interventions: Device: fixed retainer
- removable mandibular retainer (Active Comparator): Group without fixed retainer will be wearing removable thermoplastic vacuum-formed Essix retainer
  Interventions: Device: removable retainer

INTERVENTIONS:
Device: fixed retainer — bonded lingual mandibular fixed retainer on frontal teeth 33-43
  Arms: fixed mandibular lingual rectangular retainer 0.673 x 0.268 mm; fixed mandibular lingual round retainer 0.40 mm
Device: removable retainer — thermoplastic vacuum-formed removable mandibular retainer
  Arms: removable mandibular retainer

SUMMARY:
Objective is to assess changes of dentition and periodontium, and hygiene in retention after the end of the active phase of orthodontic treatment, and relationship with gender, type of retention appliance, pre-therapeutic condition of dentition and duration of active phase of treatment.

DETAILED DESCRIPTION:
A total of 152 subjects will be recruited and randomly assigned into three groups. First group will have a square 8-stranded 0.673x0.268 mm retainer wire bonded in mandibular teeth after completing the active phase of comprehensive orthodontic treatment with fixed appliances. Retainer will be bonded on lingual site canine to canine on each tooth. Second group will have a round 6-stranded 0.40 mm retainer in mandible. Third group will be without fixed retainer, only with thermoplastic vacuum-formed removable Essix retainer in mandible.

Subjects will be examined before orthodontic treatment (T0), upon completion of treatment (T1), six months in retention (T2), two years (T3) and three years in retention (T4). Changes in intercanine width, relapse (unexpected tooth movements), retainer failure, accumulation of biofilm, calculus and gingivitis will be assessed.

ELIGIBILITY:
Inclusion Criteria: finished orthodontic treatment, participants must have all permanent teeth Exclusion Criteria: hypodontia, missing teeth

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
severity of relapse (unexpected tooth movement in mandibular frontal area) at 1 year | 1 year
  the unabbreviated scale title: Little Irregularity Index (used to measure the crowding)- numerical rating scale in millimeters the minimum and maximum values: 0,10 higher scores mean a worse outcome lower scores mean a better outcome
severity of relapse (unexpected tooth movement in mandibular frontal area) at 2 years | 2 years
  the unabbreviated scale title: Little Irregularity Index (used to measure the crowding)- numerical rating scale in millimeters the minimum and maximum values: 0,10 higher scores mean a worse outcome lower scores mean a better outcome
severity of relapse (unexpected tooth movement in mandibular frontal area) at 3 years | 3 years
  the unabbreviated scale title: Little Irregularity Index (used to measure the crowding)- numerical rating scale in millimeters the minimum and maximum values: 0,10 higher scores mean a worse outcome lower scores mean a better outcome
incidence of retainer failure (debonding, breakage) at 2 years | 2 years
  percentage of cases with at least one fixed retainer failure, the minimum and maximum values 0%,100% higher scores mean a worse outcome, lower scores mean a better result
incidence of retainer failure (debonding, breakage) at 3 years | 3 years
  percentage of cases with at least one fixed retainer failure, the minimum and maximum values 0%,100% higher scores mean a worse outcome, lower scores mean a better result
extent of biofilm accumulation at 2 years | 2 years
  the unabbreviated scale title: Silness and Loe Plaque Index-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better result
extent of biofilm accumulation at 3 years | 3 years
  the unabbreviated scale title: Silness and Loe Plaque Index-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better result

SECONDARY OUTCOMES:
incidence of intercanine width change | 3 years
  percentage of cases with intercanine width change, the minimum and maximum values 0%,100% higher scores mean a worse outcome, lower scores mean a better result
changes of intercanine width | 2 years, 3 years
  the unabbreviated scale title: intercanine width change in millimeters, the minimum and maximum values 0,5, higher scores mean a worse outcome, lower result mean a better outcome
extent of calculus accumulation at 2 years | 2 years
  the unabbreviated scale title: Calculus Surface Index (CSI)-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better outcome
extent of calculus accumulation at 3 years | 3 years
  the unabbreviated scale title: Calculus Surface Index (CSI)-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better outcome

OTHER OUTCOMES:
incidence of relapse at 2 years | 2 years
  the unabbreviated scale title: percentage of relapsed cases; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better outcome
incidence of relapse at 3 years | 3 years
  the unabbreviated scale title: percentage of relapsed cases; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better outcome
extent of gingivitis at 2 years | 2 years
  the unabbreviated scale title: Bleeding on probing (BOP)-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better result
extent of gingivitis at 3 years | 3 years
  the unabbreviated scale title: Bleeding on probing (BOP)-ratio of measuring sites in mandibular central sextant; the minimum and maximum values 0%,100%, higher scores mean a worse outcome, lower scores mean a better result
duration of orthodontic treatment in months | 1 year
  the unabbreviated scale title: numerical rating scale the minimum and maximum values: 0,30
satisfaction with stability of results in retention period | 3 years
  Participant's satisfaction with stability of results as assessed using a 5-point Likert scale. Scores range from "very unsatisfied" (1) to "very satisfied" (5). Higher scores mean a better outcome, lower scores mean a worse outcome
costs total | 3 years
  calculation of costs of retention: failures and new retainers in euros
loss of productivity | 3 years
  the unabbreviated scale title: number of check-ups in retention period; the minimum and maximum values 0,10; higher scores mean a worse outcome, lower scores mean a better result the minimum and maximum values: 0,30

CONTACTS AND LOCATIONS:
Overall Officials: Silvija Kanižaj Ugrin, DDM, Principal Investigator — Poliklinika Orthonova
Locations (1):
- Poliklinika Orthonova, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
on request

REFERENCES:
- [Derived] Kanizaj Ugrin S, Spalj S. Comparison of efficacy of thermoplastic retainer with round and rectangular bonded lingual wire retainer in the mandible two years after orthodontic treatment: a randomised controlled trial. Clin Oral Investig. 2024 Mar 1;28(3):183. doi: 10.1007/s00784-024-05572-y. PMID 38424224